CLINICAL TRIAL: NCT04807218
Title: Virta Intervention in CommuniTies in cOloRado (VICTOR-Pilot) Pilot Study to Improve Diabetes and Cardiovascular Risk in Rural Communities
Brief Title: Virta Intervention in CommuniTies in cOloRado (VICTOR-Pilot)
Acronym: VICTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado Prevention Center (Other)
Collaborators: Virta Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VIRT-001
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Community Health Workers; Nutritional Ketosis; Patient Navigator; Diabetes; Referral
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nutritional Ketosis Intervention Referral (Active Comparator): The comprehensive remotely-delivered continuous remote care to induce nutritional ketosis combined with remote medication management is the Virta treatment, and while on this treatment, subjects will have access to Virta health coaches and licensed medical providers who will perform medical therapy management, health coaching, nutrition and behavior change education, biometric feedback, and the option to participate in a community for peer support.
  Interventions: Behavioral: Virta Health
- CHHS Standard Care - Delayed Referral to Nutritional Ketosis Intervention (Active Comparator): All subjects will be enrolled in Colorado Heart Healthy Solutions (CHHS), which consists of community health worker (CHW) contact and sessions on: 1) cardiovascular disease knowledge; 2) Health behavior change through skill building to improve diet (e.g., portion sizes, increasing fruit/vegetable intake, reducing intake of sugar sweetened beverages, decreasing fast food meals, etc.), increase physical activity, and improve well-being, tailored to individual subjects' risk profile and self-identified goals; and 3) Connection to services including primary care, mental health services if needed, and relevant community programs to address barriers (e.g. food insecurity, need for legal help) or to promote behavior change (e.g. free/low cost exercise programs).
  Interventions: Behavioral: Virta Health

INTERVENTIONS:
Behavioral: Virta Health — The comprehensive remotely-delivered continuous remote care to induce nutritional ketosis combined with remote medication management is the Virta treatment, and while on this treatment, subjects will have access to Virta health coaches and licensed medical providers who will perform medical therapy management, health coaching, nutrition and behavior change education, biometric feedback, and the option to participate in a community for peer support.

SUMMARY:
The VICTOR study plans to include rural communities served by Colorado Heart Healthy Solutions (CHHS) program and find out whether participants will accept a referral to a comprehensive virtual lifestyle intervention, Virta Health. The Virta Health program induces nutritional ketosis to improve glucose control in individuals with type 2 diabetes. The study will inform the acceptability of the referral, the retention of participants in lifestyle intervention, and the durability of effects on glucose control after the lifestyle intervention has ended.

DETAILED DESCRIPTION:
In rural communities served by Colorado Heart Healthy Solutions (CHHS), referral to a comprehensive remotely-delivered (virtual) continuous remote care to induce nutritional ketosis combined with remote medication management will improve glycemic control in patients with type 2 diabetes as compared with standard care. The study intervention is the referral. Subjects are not mandated to receive Virta treatment and are welcome to continue in the study whether or not the referral is accepted. 2 rural communities served by CHHS have been chosen as recruitment sites. Study patients will be randomized at the site level.

Objectives

Primary: To assess glycemic control in patients with type 2 diabetes living in a rural community referred to a comprehensive remotely-delivered continuous remote care to induce nutritional ketosis combined with remote medication management (termed "continuous remote care") as compared with those living in a rural community offered standard care.

Secondary:

1. To assess the effects of referral to continuous remote care as compared with standard care on body weight and on body mass index
2. To assess the effects of referral to continuous remote care as compared with standard care on number and doses of anti-hyperglycemic medications
3. To determine the durability of a continuous remote care intervention when paired with ongoing community health worker support

   Exploratory:
4. To assess the effects of referral to continuous remote care as compared with standard care on LDL-cholesterol, fasting glucose, and fasting triglyceride/HDL-cholesterol ratio
5. To assess patient-reported outcomes of continuous remote care as compared with standard care
6. To determine enrollment rate (offered vs accepted) in patients with type 2 diabetes living in rural communities referred to continuous remote care.
7. To determine active engagement (number, timing, and types of 2-way contacts) and retention in patients with type 2 diabetes living in rural communities referred to continuous remote care.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide electronic informed consent
2. Age 18 - 79 years old
3. Type 2 diabetes mellitus diagnosis by self-report and/or medical history
4. Taking 1 or more antihyperglycemic medications
5. Current HbA1c > 7.5%
6. Body mass index (BMI) 25 kg/m2 or greater
7. Capable of engaging in virtual care

Exclusion Criteria:

1. Type 1 diabetes
2. Pregnant or planning pregnancy within the next 9 months
3. Lactating
4. Admission for diabetic ketoacidosis (DKA) or hyperglycemic hyperosmolar syndrome (HHS) within the last 12 months
5. Life expectancy <1 year
6. Postural orthostatic tachycardia syndrome (POTS) and/or recurrent syncope
7. Active severe psychiatric or medical condition(s) such as advanced renal (end-stage renal disease or CKD stage 4 or 5; eGFR <30 mL/min), cardiac (NYHA Class 4 heart failure), or hepatic dysfunction (Child-Pugh Class C)
8. Any condition which in the opinion of the investigator would make the study unsuitable for the subject including investigator opinion regarding inability to comply with Virta instructions

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c (Percent) | 3.5 months
  Change from baseline hemoglobin A1c (Percent) among patients referred to continuous remote care (Group 1) versus standard care (Group 2)

SECONDARY OUTCOMES:
Change in BMI | Baseline versus 3.5 months, 3.5 months versus 7 months, baseline versus10 months
  Among Group 1 versus Group 2 subjects, change in body mass index (kg/m2)
Change in hemoglobin A1c | 3.5 months versus 7 months, baseline versus 10 months
  Among Group 1 versus Group 2 subjects, difference in hemoglobin A1c
Change in number and/or doses of anti-hyperglycemic medications • doses of anti-hyperglycemic medications | Baseline versus 3.5 months, 3.5 months versus 7 months, baseline versus 10 months
  Among Group 1 versus Group 2 subjects, difference in:
  * number of anti-hyperglycemic medications
  * doses of anti-hyperglycemic medications

OTHER OUTCOMES:
Acceptance of referral to continuous remote care | Baseline in Group 1 versus 3.5 months in Group 2
  Proportion agreeing to participate in continuous remote care in Group 1 at baseline versus at 3.5 months in Group 2
Change in fasting triglyceride/HDL ratio | Baseline versus 3.5 months, 3.5 months versus 7 months, baseline versus 10 months
  Among Group 1 versus Group 2 subjects, change from in fasting triglyceride/HDL ratio
Change in LDL-cholesterol | Baseline versus 3.5 months, 3.5 months versus 7 months, baseline versus 10 months
  Among Group 1 versus Group 2 subjects, change from in LDL-cholesterol
Change in fasting glucose | Baseline versus 3.5 months, 3.5 months versus 7 months, baseline versus 10 months
  Among Group 1 versus Group 2 subjects, change from in fasting glucose
Acceptance/continuation of referral to continuous remote care | Baseline and 3.5 months
  Among Group 1 subjects, proportion agreeing to participate in continuous remote care
Continuation of referral in Group 1 versus acceptance of referral in Group 2 | 3.5 months
  Among Group 1 versus Group 2 subjects, proportion agreeing to participate/continue in continuous remote care
Change in perceived health status | Baseline, 3.5 months, 7 months and 10 months
  Among Group 1 and Group 2 subjects, evaluation over time (i.e. 3 months post-intervention) in perceived health status as assessed by question 1 of the Short Form Health Survey (SF-1).
Change in diabetes treatment satisfaction | Baseline, 3.5 months, 7 months and 10 months
  Among Group 1 and Group 2 subjects, evaluation over time at baseline, in diabetes treatment satisfaction as assessed by the Diabetes Treatment Satisfaction Questionnaire. The scale for the survey questions is 0-6. In general, a higher score indicates a higher level of satisfaction with diabetic treatment.
Count of 2-way contacts among subjects | 3.5 months and 7 months
  Among Group 1 and Group 2 subjects, evaluation in active engagement as assessed by number of 2-way contacts.
Acceptability of referral | Group 1: baseline, 3.5 months and 7 months / Group 2: 3.5 months and 7 months
  Among Group 1 subjects at baseline 3.5 and 7 months, and Group 2 subjects at 3.5 and 7 months. Participants will be asked 'Did you complete the referral to Virta Health?' Yes/No
Acceptability of referral over time | Group 1: baseline, 3.5 months and 7 months / Group 2: 3.5 months and 7 months
  Among Group 1 subjects at baseline 3.5 and 7 months, and Group 2 subjects at 3.5 and 7 months. Participants will be asked if they are still continuing their treatment with Virta Health.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Low Wang, MD, Principal Investigator — CPC Clinical Research
Locations (3):
- United States (3):
  - Northwest Colorado Health - Community Health Center & Prevention Services Craig, Craig, Colorado
  - High Plains Community Health Center, Lamar, Colorado
  - Chaffee County Public and Environmental Health, Salida, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yaemsiri S, Alfier JM, Moy E, Rossen LM, Bastian B, Bolin J, Ferdinand AO, Callaghan T, Heron M. Healthy People 2020: Rural Areas Lag In Achieving Targets For Major Causes Of Death. Health Aff (Millwood). 2019 Dec;38(12):2027-2031. doi: 10.1377/hlthaff.2019.00915. PMID 31794308
- [Background] American Diabetes Association. 1. Improving Care and Promoting Health in Populations: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S7-S14. doi: 10.2337/dc21-S001. PMID 33298412
- [Background] Lee JY, Lee SWH. Telemedicine Cost-Effectiveness for Diabetes Management: A Systematic Review. Diabetes Technol Ther. 2018 Jul;20(7):492-500. doi: 10.1089/dia.2018.0098. Epub 2018 May 29. PMID 29812965
- [Background] McKenzie AL, Hallberg SJ, Creighton BC, Volk BM, Link TM, Abner MK, Glon RM, McCarter JP, Volek JS, Phinney SD. A Novel Intervention Including Individualized Nutritional Recommendations Reduces Hemoglobin A1c Level, Medication Use, and Weight in Type 2 Diabetes. JMIR Diabetes. 2017 Mar 7;2(1):e5. doi: 10.2196/diabetes.6981. PMID 30291062
- [Background] Bhanpuri NH, Hallberg SJ, Williams PT, McKenzie AL, Ballard KD, Campbell WW, McCarter JP, Phinney SD, Volek JS. Cardiovascular disease risk factor responses to a type 2 diabetes care model including nutritional ketosis induced by sustained carbohydrate restriction at 1 year: an open label, non-randomized, controlled study. Cardiovasc Diabetol. 2018 May 1;17(1):56. doi: 10.1186/s12933-018-0698-8. PMID 29712560
- [Background] Hallberg SJ, McKenzie AL, Williams PT, Bhanpuri NH, Peters AL, Campbell WW, Hazbun TL, Volk BM, McCarter JP, Phinney SD, Volek JS. Author Correction: Effectiveness and Safety of a Novel Care Model for the Management of Type 2 Diabetes at 1 Year: An Open-Label, Non-Randomized, Controlled Study. Diabetes Ther. 2018 Apr;9(2):613-621. doi: 10.1007/s13300-018-0386-4. PMID 29508274
- [Background] Krantz MJ, Coronel SM, Whitley EM, Dale R, Yost J, Estacio RO. Effectiveness of a community health worker cardiovascular risk reduction program in public health and health care settings. Am J Public Health. 2013 Jan;103(1):e19-27. doi: 10.2105/AJPH.2012.301068. Epub 2012 Nov 15. PMID 23153152
- [Background] Centers for Disease Control and Prevention. Diabetes Basics: Type 2 diabetes. Page last reviewed: May 30, 2019. https://www.cdc.gov/diabetes/basics/type2.html. Accessed 06 January 2021.
- [Background] Kazemian P, Shebl FM, McCann N, Walensky RP, Wexler DJ. Evaluation of the Cascade of Diabetes Care in the United States, 2005-2016. JAMA Intern Med. 2019 Oct 1;179(10):1376-1385. doi: 10.1001/jamainternmed.2019.2396. PMID 31403657
- [Background] Stellefson M, Dipnarine K, Stopka C. The chronic care model and diabetes management in US primary care settings: a systematic review. Prev Chronic Dis. 2013;10:E26. doi: 10.5888/pcd10.120180. PMID 23428085
- [Background] Egbujie BA, Delobelle PA, Levitt N, Puoane T, Sanders D, van Wyk B. Role of community health workers in type 2 diabetes mellitus self-management: A scoping review. PLoS One. 2018 Jun 1;13(6):e0198424. doi: 10.1371/journal.pone.0198424. eCollection 2018. PMID 29856846
- [Background] Understanding Scope and Competencies: A Contemporary Look at the United States Community Health Worker Field: Progress Report of the Community Health Worker (CHW) Core Consensus (C3) Project: Building National Consensus on CHW Core Roles, Skills, and Qualities [Internet], 2016. Available from: http://files.ctctcdn.com/a907c850501/1c1289f0-88cc-49c3-a238-66def942c147.pdf. Accessed 04 November 2020.
- [Background] Lee SWH, Chan CKY, Chua SS, Chaiyakunapruk N. Comparative effectiveness of telemedicine strategies on type 2 diabetes management: A systematic review and network meta-analysis. Sci Rep. 2017 Oct 4;7(1):12680. doi: 10.1038/s41598-017-12987-z. PMID 28978949
- [Background] Faruque LI, Wiebe N, Ehteshami-Afshar A, Liu Y, Dianati-Maleki N, Hemmelgarn BR, Manns BJ, Tonelli M; Alberta Kidney Disease Network. Effect of telemedicine on glycated hemoglobin in diabetes: a systematic review and meta-analysis of randomized trials. CMAJ. 2017 Mar 6;189(9):E341-E364. doi: 10.1503/cmaj.150885. Epub 2016 Oct 31. PMID 27799615
- [Background] Marcolino MS, Maia JX, Alkmim MB, Boersma E, Ribeiro AL. Telemedicine application in the care of diabetes patients: systematic review and meta-analysis. PLoS One. 2013 Nov 8;8(11):e79246. doi: 10.1371/journal.pone.0079246. eCollection 2013. PMID 24250826
- [Background] American Diabetes Association. 5. Facilitating Behavior Change and Well-being to Improve Health Outcomes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S53-S72. doi: 10.2337/dc21-S005. PMID 33298416
- [Background] Sainsbury E, Kizirian NV, Partridge SR, Gill T, Colagiuri S, Gibson AA. Effect of dietary carbohydrate restriction on glycemic control in adults with diabetes: A systematic review and meta-analysis. Diabetes Res Clin Pract. 2018 May;139:239-252. doi: 10.1016/j.diabres.2018.02.026. Epub 2018 Mar 6. PMID 29522789
- [Background] Snorgaard O, Poulsen GM, Andersen HK, Astrup A. Systematic review and meta-analysis of dietary carbohydrate restriction in patients with type 2 diabetes. BMJ Open Diabetes Res Care. 2017 Feb 23;5(1):e000354. doi: 10.1136/bmjdrc-2016-000354. eCollection 2017. PMID 28316796
- [Background] Athinarayanan SJ, Adams RN, Hallberg SJ, McKenzie AL, Bhanpuri NH, Campbell WW, Volek JS, Phinney SD, McCarter JP. Long-Term Effects of a Novel Continuous Remote Care Intervention Including Nutritional Ketosis for the Management of Type 2 Diabetes: A 2-Year Non-randomized Clinical Trial. Front Endocrinol (Lausanne). 2019 Jun 5;10:348. doi: 10.3389/fendo.2019.00348. eCollection 2019. PMID 31231311
- [Background] Senn S. Crossover Trials in Clinical Research. (1993) John Wiley & Sons, New York.
- [Background] Littell RC, et al. SASA System for Linear Models. (1991) Third edition, Cary, NC. SAS Institute, Inc.
- [Background] United States Food and Drug Administration. E6(R2) Good Clinical Practice: Integrated Addendum to ICH E6(R1). Guidance for Industry. OMB Control No. 0910-0843. March, 2018